CLINICAL TRIAL: NCT01126385
Title: A Prospective Case Series to Evaluate Handling and Feasibility of DensiProbe Spine Assessing Vertebral Bone Strength in Patients Undergoing Transpedicular Fixation of the Spine - a Pilot Study
Brief Title: Pilot Study to Evaluate Feasibility of DensiProbe Spine Assessing Bone Strength in Spinal Surgery
Acronym: DensiProbe
Status: Completed | Type: Observational
Sponsor: AO Clinical Investigation and Publishing Documentation (Other)
Collaborators: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Organization: AO Innovation Translation Center (Other)
Other Study IDs: DensiProbe Spine 2010
Record Dates: First submitted 2010-05-18; First posted 2010-05-19 (Estimated); Last update posted 2013-01-25 (Estimated); Status verified 2013-01

CONDITIONS: Spinal Diseases
Keywords: Spinal Diseases; Bone strength; Transpedicular fixation; Dorsal instrumentation; DensiProbe
MeSH Terms: conditions — Spinal Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Transpedicular stabilization: Patients undergoing transpedicular stabilization of the spine
  Interventions: Device: DensiProbe Spine

INTERVENTIONS:
Device: DensiProbe Spine — Intraoperative DensiProbe Spine measurements

SUMMARY:
A new mechanical device was developed in order to provide the surgeon with intraoperative information about the mechanical strength of the cancellous bone within the vertebral body. DensiProbe Spine is intended to be used in patients undergoing transpedicular stabilization of the thoracolumbar spine. The objective of the DensiProbe Spine pilot study is to investigate the handling and feasibility of the DensiProbe Spine measurement device.

DETAILED DESCRIPTION:
Osteoporotic fragility fractures often occur in the spine. A common surgical technique is the transpedicular fixation using pedicle screws. A major complication of this treatment is a cut-out or back-out of the screw due to insufficient anchorage of the implant in the vertebral body.

A new mechanical device was developed in order to provide the surgeon with intraoperative information about the mechanical strength of the cancellous bone. In cases of low bone quality, the treatment can be adapted to the patient's condition, for example by augmentation of the screw anchorage using bone cement. However, this treatment involves a risk of cement leakage and subsequent pulmonary embolism or nerve damage. Furthermore, cement augmentation is time-consuming. Therefore, there is a need for a diagnostic device that can intraoperatively support the surgeon's decision on the appropriate treatment.

DensiProbe Spine was developed accordingly to the clinically approved DensiProbe Hip, which was designed for the same diagnostic reasons in patients with hip fractures undergoing fracture fixation with the dynamic hip screw (DHS). However, the application of bone strength measurements in the spine is in so far different to the hip as the anatomical dimensions in the spine are much smaller and lower values of bone mineral density (BMD) and bone strength are expected.

The objective of this pilot study is to investigate the handling and feasibility of the newly developed DensiProbe Spine measurement device. In case of a positive result of the pilot study, a multicenter cohort study will be performed in order to clinically validate the DensiProbe Spine device by assessing the correlation between DensiProbe Spine measurements and the amounts of pedicle screw migration in patients undergoing transpedicular fixation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Indication for transpedicular fixation of the thoracolumbar spine
* Ability to understand and read local language at an elementary level
* Signed informed consent by patient or legal guardian to participate in the study according to the protocol

Exclusion Criteria:

* Patients who are legally incompetent
* Scoliosis (Cobb angle on AP radiograph > 10°)
* Benign or malign vertebral bone tumour
* Active malignancy
* Infection diseases, eg. hepatitis, human immunodeficiency virus (HIV)
* Pre-drilling with power-drill
* Life-threatening condition
* Drug or alcohol abuse
* Participation in any other medical device or drug study that could influence the results of the present study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing transpedicular stabilization of the spine
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2010-08; Primary Completion 2012-03 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Surgeon's compliance- and handling-oriented questionnaire | Baseline
  The general satisfaction of the surgeon with DensiProbe Spine as well as specific problems that are likely to occur during the measurement with DensiProbe Spine will be assessed
Intra- and post-operative adverse events | Up to 2 months postsurgery
  All intra- and postoperative adverse events will be assessed and analyzed regarding their relationship to the study device

SECONDARY OUTCOMES:
Bone mineral density | Baseline
  The bone mineral density will be measured preoperatively in the lumbar spine (L1-L4) using DXA in order to assess local bone status.
Pedicle screw migration | 2 months postsurgery
  The migration of the pedicle screw will be performed by measuring the angle between the pedicle screw axis and the caudal endplate. The amount of screw migration is defined as the difference in that angle between the baseline (postoperative) and the two month lateral x-rays
QCT analysis of bone biopsies | Baseline
  For each vertebral body under investigation a probe of trabecular bone is obtained to determine bone quality using quantitative micro-CT analysis
Application of bone cement | Baseline
  For each patient the surgeon decides whether or not augmentation with bone cement is necessary

CONTACTS AND LOCATIONS:
Overall Officials: Lorin M Benneker, MD, Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (2):
- Switzerland (2):
  - Klinik Sonnenhof, Bern, Canton of Bern
  - Inselspital, Bern, Canton of Bern